CLINICAL TRIAL: NCT02008747
Title: Effects of Prophylactic Administration of Magnesium Sulfate on the Incidence of Atrial Fibrillation and Chronic Neuropathic Pain After Thoracotomy for Lung Resection.
Brief Title: Atrial Fibrillation and Neuropathic Pain After Thoracotomy and Continuous Application of Magnesium Sulphate.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSK 002
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Atrial Fibrillation; Neuropathic Pain
Keywords: Atrial fibrillation; Neuropathic pain; Posterolateral thoracotomy; Lung resection
MeSH Terms: conditions — Atrial Fibrillation; Neuralgia | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulphate (Active Comparator): The patients in this group underwent general anaesthesia with total intravenous anesthesia containing Remifentanyl (0,3 mg/kg ideal body weight/h), Propofol (4 mg/kg ideal body weight/h) and Atracurium.
  They also received 40mg/kg ideal body weight magnesium sulphate by bolus injection before the operation started, followed by a continuous application of 10mg/kg ideal body weight/hour for 24 hours.
  Interventions: Drug: Magnesium sulphate
- No treatment (No Intervention): The patients in this group underwent general anaesthesia with total intravenous anesthesia containing Remifentanyl (0,3 mg/kg ideal body weight/h), Propofol (4 mg/kg ideal body weight/h) and Atracurium. They received no additional medication.

INTERVENTIONS:
Drug: Magnesium sulphate — Continuous application of magnesium sulphate applied 40 mg/kg ideal body weight by bolus before the operation started, followed by a continuous infusion of 10 mg/kg ideal body weight/h for 24 hours
  Other Names: Mg 5 Sulfat 10%
  Arms: Magnesium sulphate

SUMMARY:
Atrial fibrillation and chronic neuropathic pain are adverse events occurring after posterolateral thoracotomy for lung resection. The continuous application of magnesium sulphate may have a prophylactic effect. The investigators record the incidence of atrial fibrillation during a seven day period after thoracotomy as well as the incidence of chronic neuropathic pain during a three months period, comparing one group with a continuous application of magnesium sulphate against one group without magnesium sulphate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* posterolateral thoracotomy for lung parenchyma resection
* informed consent

Exclusion Criteria:

* hypersensitivity for magnesium sulphate
* pre-existing atrial fibrillation
* participation in another trial
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation | Up to 168 hours after operation
  The incidence of atrial fibrillation was recorded using a 12 lead ECG for a period of 7 days after operation

SECONDARY OUTCOMES:
Chronic neuropathic pain | Three months
  The incidence of neuropathic pain was recorded using the LANSS Score during a period of three months after posterolateral thoracotomy for lung resection.

OTHER OUTCOMES:
Hypotonia | 24 hours perioperative
  The incidence of hypotonia during the time of continuous magnesium sulphate application was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Grietje Beck, Prof., Study Chair — HSK Wiesbaden
Locations (1):
- HSK, Wiesbaden, Germany